CLINICAL TRIAL: NCT02313285
Title: An Open-label, Long-term Follow-up Study Of Multiple Sclerosis Patients Who Participated In Genzyme-sponsored Studies of GZ402668
Brief Title: A Long-term Follow-up Study Of Multiple Sclerosis Patients Who Participated In Genzyme-sponsored Studies of GZ402668
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: LTS14120; 2014-001592-31 (EudraCT Number); U1111-1158-9815 (Other: UTN)
Record Dates: First submitted 2014-12-04; First posted 2014-12-10 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GZ402668: Patient who received GZ402668 in prior study (TDU13475 or TDU14981)
- Placebo: Patient who received placebo in prior study (TDU13475 or TDU14981)

SUMMARY:
Primary Objective:

To assess the long-term safety of GZ402668 in patients with multiple sclerosis (MS) who received prior treatment during the TDU13475 or TDU14981 studies.

Secondary Objectives:

To assess the pharmacokinetics of GZ402668 in patients with MS. To assess the pharmacodynamics of GZ402668 in patients with MS. To assess the immunogenicity of GZ402668 in patients with MS.

DETAILED DESCRIPTION:
The total study duration for a patient is approximately 47 months.

There is no administration of GZ402668 in the LTS14120 study. Patients who already received investigational medicinal product (GZ402668 or placebo) in TDU13475 or TDU14981 will be followed up to 47 months in the LTS14120.

Note: Patients from TDU14981 study (sanofi-sponsored) will participate in LTS14120 study. In order to keep consistent among all study related documents, the title of the LTS14120 study is not amended.

ELIGIBILITY:
Inclusion criteria:

Received investigational medicinal product (GZ402668 or placebo) in TDU13475 or TDU14981

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received study drug in the clinical study TDU13475
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 4 years
Safety, as assessed by clinical (physical examination), laboratory (hematology, creatinine, and urinalysis with microscopy), ECG, and vital sign events | monthly for up to 4 years
Clinically significant changes in thyroid function tests from baseline | every 3 months for 4 years

SECONDARY OUTCOMES:
Time to lymphocyte repopulation | 4 years
Number of patients with anti-drug antibodies | monthly for first 3 months then at 6 and 12 months for first 1 year
Serum concentrations of GZ402668 | monthly for first 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Albach FN, Geier C, Keicher C, Posch MG, Schreiber SJ, Grutz G, Akyuz L, Luo X, Le-Halpere A, Truffinet P, Wagner F. Phase 1 Trials of Gatralimab, a Next-Generation Humanized Anti-CD52 Monoclonal Antibody, in Participants with Progressive Multiple Sclerosis. Neurol Ther. 2024 Dec;13(6):1607-1625. doi: 10.1007/s40120-024-00659-w. Epub 2024 Sep 9. PMID 39251561